CLINICAL TRIAL: NCT06149650
Title: Chronic Limb-Threatening Ischemia Treated With Intravascular Lithotripsy Observational Study
Acronym: CALCIO
Status: Recruiting | Type: Observational
Sponsor: Cardiovascular and Interventional Radiological Society of Europe (Other)
Collaborators: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CALCIO
Record Dates: First submitted 2023-11-15; First posted 2023-11-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Chronic Limb-Threatening Ischemia
Keywords: CLTI
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Full cohort: Intravascular lithotripsy of femoropopliteal and crural lesions as per standard of care
  Interventions: Device: Shockwave Medical IVL System

INTERVENTIONS:
Device: Shockwave Medical IVL System — Comprehensive system consisting of generator, a connector cable and a single-use sterile catheter with integrated balloon for intravascular lithotripsy of peripheral artery calcification.

SUMMARY:
CALCIO is a multicentre, prospective, observational cohort study that will collect real world data on the use of intravascular Lithotripsy (IVL) with the Shockwave IVL system to disrupt calcified femoropopliteal and crural lesions in patients with chronic limb-threatening ischemia (CLTI). The primary objective of CALCIO is to understand the effectiveness of IVL in promoting wound healing and preventing amputation. The secondary objectives of CALCIO are to evaluate the immediate effectiveness of the treatment in restoring vessel patency as well as its safety and impact on patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic limb-threatening ischemia (Rutherford Category ≥4)
* Femoropopliteal and/or crural calcified lesions visible on fluoroscopy;
* Treatment with IVl using the Shockwave Medical IVL System.

Exclusion Criteria:

* < 18 years old;
* Incapacity or refusal to give informed consent;
* Ongoing pregnancy;
* Endovascular procedure(s) on the treatment site within 4 weeks before the planned IVL treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CLTI patients with calcified femoropopliteal or crural lesions visible on fluoroscopy and treated with Intravascular Lithotripsy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2028-07-15 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Wound healing and freedom from amputation | 12 months
  Composite of wound healing defined as the healing status of the dominant ischemic wound of the target limb (complete, partial, unchanged, worsening) and freedom from amputation defined as the absence of any amputation of the treated limb: minor (digital, metatarsal), major below the knee or major above the knee (excluding any amputation planned before the IVL procedure).

SECONDARY OUTCOMES:
Wound healing | 24 months
  Healing status of the dominant ischemic wound of the target limb (complete, partial, unchanged, worsening)
Freedom from amputation | 24 months
  Absence of any amputation of the treated limb: minor (digital, metatarsal), major below the knee or major above the knee (excluding any amputation planned before the IVL procedure).
Amputation-free survival | through study completion, approximately 2 years
  time between IVL treatment and amputation of the target limb, minor (digital, metatarsal), major below the knee or major above the knee (excluding any amputation planned before the IVL procedure)
Change in Rutherford classification category | 12 and 24 months
  Seven classification categories, from 0 (asymptomatic) to 6 (Major tissue loss)
Change in foot ischemia | 12 and 24 months
  Change in ankle-brachial index or toe pressure, depending on which data is available
Change in WIfi score | 12 and 24 months
  Three-digit score for comprehensive assessment of wound, ischemia and foot infection
Freedom from clinically-driven target lesion revascularization (CD-TLR) | 12 and 24 months
  freedom from any endovascular re-intervention to the target lesion (± 10 mm) or surgical bypass performed because of restenosis or occlusion of the target lesion.
CD-TLR-free survival | through study completion, approximately 2 years
  time between IVL treatment and any endovascular re-intervention to the target lesion (± 10 mm)
Primary patency rate | 12 and 24 months
  freedom from total occlusion without any endovascular or surgical re-intervention to the target lesion (± 10 mm)
Assisted primary patency rate | 12 and 24 months
  freedom from total occlusion following additional endovascular or surgical intervention(s) due to restenosis of the target lesion
Secondary patency rate | 12 and 24 months
  freedom from total occlusion following additional endovascular or surgical intervention(s) due to occlusion of the target lesion
Technical success of IVL | on the day of the procedure
  residual diameter stenosis ≤30% after IVL and before any potential adjunctive intervention
Overall procedural success | on the day of the procedure
  residual stenosis ≤30% by the end of the complete procedure
Frequency and severity of procedural complications and other adverse events | Within 30 days after the procedure
  Grading according to the classification system of the Cardiovascular and Interventional Radiological Society of Europe
Patient-reported health-related quality-of-life | at 6, 12 and 24 months
  EuroQol questionnaire EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Raman Uberoi, Dr, Study Chair — Oxford University Hospital NHS Foundation Trust, Oxford, United Kingdom; Christoph Binkert, Prof. Dr, Study Chair — Cantonal Hospital Winterthur, Winterthur, Switzerland; Peter Reimer, Prof. Dr, Study Chair — Municipal Clinic Karlsruhe, Karlsruhe, Germany
Locations (39):
- Austria (5):
  - Krankenhaus der Barmherzigen Brüder, Eisenstadt
  - Medizinische Universität Graz, Graz
  - Krankenhaus Barmherzige Brüder Linz, Linz
  - Klinik Hietzing, Vienna
  - Klinik Florisdorf, Vienna
- Hôpital Sacré Coeur de Montréal, Montreal, Canada
- France (3):
  - CHU François Mitterrand, Dijon
  - Institute Mutualiste Montsouris, Paris
  - Rhéna Clinique de Strasbourg, Strasbourg
- Germany (10):
  - Universitätsklinikum Köln, Cologne
  - Universitätsmedizin Essen, Essen
  - KRH Klinikum Robert Koch Gehrden, Hanover
  - SLK-Heilbronn, Heilbronn
  - Städtisches Klinikum, Karlsruhe
  - Evangelisches Krankenhaus, Mülheim
  - Friedrich Ebert Krankenhaus, Neumünster
  - Schön Klinik Rendsburg, Rendsburg
  - St Marien-Krankenhaus, Siegen
  - Universitätsklinikum Tübingen, Tübingen
- Semmelweis University, Budapest, Hungary
- Spain (3):
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital General de Granollers, Granollers
  - University of Navarra, Pamplona
- Switzerland (2):
  - Ente Ospedaliero Cantonale, Lugano
  - Kantonsspital Winterthur, Winterthur
- United Kingdom (14):
  - Bedfordshire Hospitals NHS Foundation Trust, Bedford
  - Frimley Health NHS Foundation Trust, Frimley
  - Hull University Teaching Hospitals NHS Trust, Hull
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - University College London Hospitals NHS Foundation Trust, London
  - Royal Free London NHS Foundation Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Sheffield Teaching Hospitals NHS FT, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Filippiadis DK, Binkert C, Pellerin O, Hoffmann RT, Krajina A, Pereira PL. Cirse Quality Assurance Document and Standards for Classification of Complications: The Cirse Classification System. Cardiovasc Intervent Radiol. 2017 Aug;40(8):1141-1146. doi: 10.1007/s00270-017-1703-4. Epub 2017 Jun 5. PMID 28584945